CLINICAL TRIAL: NCT06194240
Title: Development of an E-program to Improve the Quality of Life of People With Diabetes Based on Acceptance and Commitment Therapy (ACT)
Brief Title: Contributions of Health Psychology to Support Patients With Diabetes Through Online Tools
Acronym: DiabACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lorraine (Other)
Responsible Party: Principal Investigator, Coline Hehn, Principal investigator, University of Lorraine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: ULFFD
Record Dates: First submitted 2023-12-05; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Slow ACT (Experimental): This group will follow an intervention online based on Acceptance and Commitment Therapy (ACT).
  Interventions: Behavioral: DiabACT
- Slow Diabète (Experimental): This group will follow an online Slow Diabète (Slow Diabetes) program created by the French Federation of Diabetics.
  Interventions: Behavioral: DiabACT
- No program (No Intervention): This group will not follow an online program, in order to do the comparaison.

INTERVENTIONS:
Behavioral: DiabACT — E-program proposed to diabetic patients based on ACT therapy.
  Arms: Slow ACT; Slow Diabète

SUMMARY:
With over 4 million people living with diabetes in France, i.e. 6% of the general population, it is necessary to consider both their physical and mental health. Indeed, recent studies have shown that with a good quality of life, patients have better disease management, improved physical health and social life, and reduced anxiety and depressive symptoms.

Quality of life is at the heart of this research project. In order to improve it, several psychotherapies can be used, notably those that include mindfulness. Of all those proposed in the literature, Acceptance and Commitment Therapy (ACT), developed by Hayes, appears to be ideally suited to this objective. The aim of this psychotherapy is to improve the patient's psychological flexibility. According to the scientific literature, ACT therapy has been shown to improve the quality of life of patients living with diabetes, as well as their ability to manage their condition and reduce anxiety and depressive symptoms.

This research project aims to:

1. To help patients cope better with their illness through learning the different dimensions of ACT therapy in order to obtain a toolbox to use on a daily basis, when necessary.
2. To offer professionals alternatives to the traditional care of diabetic patients with the toolbox cited above.
3. To enable health authorities to take advantage of this program and these different exercises to reduce complications in the medium and long term for people with diabetes and change health behaviors.

In 2020, the French Diabetics Federation created the "Slow Diabetes" movement. The initial objective of which was to help people with diabetes to better cope with their isolation linked to the Covid-19 pandemic. Since its launch, this movement has taken the form of several programs lasting three or six weeks and developed to improve the general well-being of people with diabetes.

The research proposed here seeks to improve the quality of life of diabetic patients through online ACT therapy, based on the "Slow Diabetes" model.

DETAILED DESCRIPTION:
The aim of this detailed description is to present the research protocol of a controlled randomized trial to evaluate the impact of an e-program based on Acceptance and Commitment Therapy (ACT) for people living with diabetes in France on the quality of life and the psychological flexibility.

The recruitment of participants is done through a call for participation launched by the French Federation of Diabetics, during which patients have access to a Patient Information Notice (PIN) presenting the project. This PIN enable diabetic patients to find out about the different possible groups of the study and the planned randomization. In this way, they will know that they can belong to three different groups : 1) The "Slow ACT" intervention group, which will follow an intervention based on acceptance and commitment therapy (duration 6 weeks); 2) The "Slow Diabetes" control group, which will follow a Slow Diabète Summer program (duration 5 weeks - launched by the French Federation of Diabetics); 3) The "No program" control group, which will not follow either of the two interventions, and will be able to compare the data from the two groups presented above.

Finally, 15 of the people in the ACT intervention group were voluntarily recruited to a Single Case protocol. This took place over 14 weeks, with 14 measures (psychological flexibility and quality of life).

The content of the e-program ACT in which not all patients have participated is sent to all of the participants of the study at the end of it, for reasons of ethics and fairness.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be aged 18 and over,
* To live with type 1 diabetes (T1D) or type 2 diabetes (T2D),
* Be French,
* Living in France
* Understand and accept the constraints of the study,
* Have given their consent after having read the terms of the study,
* Be affiliated to social security.

Exclusion Criteria:

* Lack of autonomy making it impossible to complete the online questionnaire,
* Members of the "Slow Diabetes" group cannot have benefited from the "Slow ACT" program,
* Persons deprived of their rights, persons under guardianship.

Age, type of diabetes or gender are not inclusion criteria, but will be controlled for in the statistical analyses, along with other socio-demographic variables (i.e. level of education, socio-economic level).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
12-Item Short Form Health Survey | Before the intervention and six weeks after (when the program is finished)
  Quality of life. The minimum score is 0 (bad quality of life) and the maximum score is 100 (good quality of life).

SECONDARY OUTCOMES:
Multidimensional Psychological Flexibility Inventory | Before the intervention and six weeks after (when the program is finished)
  Psychological Flexibility. This scale is divided into twelve categories, based on functional and dysfunctional processes. For functional processes, the closer the average score is to 7, the more correct is the participant's process. On the other hand, for dysfunctional processes, if the average score is close to 7, then the process is truly dysfunctional.
Hospital Anxiety and Depression Scale | Before and after the intervention
  Anxiety and Depression. The total score ranges from 0 to 21 for each category (depression or anxiety). A score of 10 or more indicates definite symptomatology.
Basic Psychological Need Satisfaction and Frustration Scale | Before the intervention and six weeks after (when the program is finished)
  Basic psychological needs. The score is divided into six categories, according to the satisfaction or frustration of one of the three basic psychological needs. When it comes to satisfaction, the closer the score is to seven, the better it is. If the score is close to seven for frustration items, then the latter will be high.
Treatment Self-Regulation Questionnaire | Before the intervention and six weeks after (when the program is finished)
  Motivation towards treatments. Two scores are given for this 19-item scale. One for autonomous motivation, with average scores ranging from 0 (no autonomous motivation) to 7 (strong autonomous motivation) with 8 items. And another for controlled motivation, with average scores ranging from 0 (no controlled motivation) to 7 (high controlled motivation) on 11 items.
Diabetes Acceptance | Before the intervention and six weeks after (when the program is finished)
  Diabetes Acceptance and Action Scale - revised. The scale is a 9-point measure of diabetes acceptance. It is based on a five-point Likert scale ranging from never true (0) to always true (4). Higher scores mean greater acceptance and greater ability to adapt to diabetes.
Generic Adherence Profile for Chronic Diseases | Before the intervention and six weeks after (when the program is finished)
  Therapeutic adherence. The questionnaire consists of 32 items covering three components of health adherence: medication and/or medical adherence, lifestyle adherence and diet adherence. Some items measure non-adherence to therapy (items 2 and 6 to 16) and others measure adherence to therapy. Responses to the items were rated on a 4-point Likert-type scale (1, never, to 4, all the time).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - University of Lorraine, Metz
  - French Federation of Diabetics, Paris

IPD SHARING:
Plan to Share IPD: No